CLINICAL TRIAL: NCT04346472
Title: Retrospective Longitudinal Follow-up in Patients With Diffuse Low-grade Glioma With Multimodal MRI Assessment
Brief Title: Longitudinal MRI Assessment in Patients With Diffuse Low-grade Gliomas
Acronym: SPECIFY
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF9647
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Low-grade Glioma
Keywords: Glioma; Magnetic Resonance Imaging; Magnetic Resonance Angiography; Disease Progression; Supratentorial Neoplasms; Blood Volume; Contrast Media; Gadolinium DTPA; Image Processing, Computer-Assisted; Neovascularization, Pathologic; Diffuse low grade glioma; Relative regional cerebral blood volume ( rRCBV); Early prognosis of anaplasic transformation; Diffuse low grade glioma anaplasic transformation
MeSH Terms: conditions — Glioma; Disease Progression; Supratentorial Neoplasms; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gliomes de grade II initial: Gliomes de grade II initial
  Interventions: Other: Repeated Measurements of the relative regional cerebral blood volume

INTERVENTIONS:
Other: Repeated Measurements of the relative regional cerebral blood volume — Repeated Measurements of the relative regional cerebral blood volume variation through an every 6 monts Magnetic Resonance Imaging use.

SUMMARY:
Retrospective longitudinal follow-up in patients with diffuse low-grade glioma with multimodal MRI assessment

ELIGIBILITY:
Inclusion criteria:

* Initial WHO grade II
* At least 3 exploitable MRI each including a morphologic FLAIR sequence and perfusion imaging

Exclusion criteria:

-Major protected person ( trusteeship, curatorship, justice safeguard)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diffuse low-grade glioma (WHO grade II)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Longitudinal variation of the relative regional cerebral blood volume | 1 day
  Longitudinal variation of the relative regional cerebral blood volume from first pass perfusion imaging data for each MRI performed

SECONDARY OUTCOMES:
Collection of histological | 1 day
  Collection of histological
Collection of radiological | 1 day
  Collection of radiological
Collection of clinical varaibles | 1 day
  Collection of clinical varaibles

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MENJOT DE CHAMPFLEUR, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC